CLINICAL TRIAL: NCT03925129
Title: A Randomized, Placebo Controlled Trial of Transcutaneous Electrical Nerve Stimulation (TENS) for Pain Management With Medication Abortion Through 70 Days' Gestation
Brief Title: Transcutaneous Electrical Nerve Stimulation (TENS) for Pain Management With Medication Abortion Through 70 Days' Gestation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Planned Parenthood of Greater New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: TENS MAB
Record Dates: First submitted 2019-04-19; First posted 2019-04-24 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Abortion in First Trimester

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TENS (Experimental)
  Interventions: Device: high frequency TENS treatment
- Sham TENS (Sham Comparator)
  Interventions: Device: Sham TENS treatment

INTERVENTIONS:
Device: high frequency TENS treatment — Treatment with high frequency for minimum of 1 hour after misoprostol administration
  Arms: TENS
Device: Sham TENS treatment — Treatment with sham TENS device for minimum of 1 hour after misoprostol administration
  Arms: Sham TENS

SUMMARY:
This is a double-blinded, randomized, placebo-controlled trial evaluating the use of High-frequency Transcutaneous Electrical Nerve Stimulation (HfTENS) compared to sham TENS for pain control during medication abortion with mifepristone and misoprostol through 70 days' gestation.

ELIGIBILITY:
Inclusion Criteria:

* Patients seeking medication abortion with a definite, singleton, intrauterine pregnancy (IUP) < 70 days' gestation on ultrasound
* Rapid Estimate of Adult Literacy in Medicine-Short Form (REALM-SF)22 score > 4
* Age equal to or greater than 18 years
* Provide informed consent to participate
* Willing to adhere to study procedures, including access to a smart phone, ability to receive text messages and answer online surveys on smart phone

Exclusion Criteria:

* Contraindication to medication abortion
* Allergy to mifepristone or misoprostol
* Contraindication or allergy to ibuprofen
* History of cardiac arrhythmia
* Presence of an implantable device with electrical discharge, i.e. cardiac pacemaker
* History of chronic pain disorder
* Any opioid use during previous 30 days
* Current or prior use of TENS
* BMI > 30

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Pain on numeric rating scale | 8 hours following misoprostol
  Maximum pain score on an 11-point numeric rating scale, where 0 is no pain, and 10 is the worst pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ariella Goldman, MD, Principal Investigator — Planned Parenthood of Greater New York
Locations (1):
- Planned Parenthood of New York City - Margaret Sanger Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goldman AR, Porsch L, Hintermeister A, Dragoman M. Transcutaneous Electrical Nerve Stimulation to Reduce Pain With Medication Abortion: A Randomized Controlled Trial. Obstet Gynecol. 2021 Jan 1;137(1):100-107. doi: 10.1097/AOG.0000000000004208. PMID 33278292